CLINICAL TRIAL: NCT06657599
Title: Malnutrition is a Severe Health Issue for Cancer Patients. This Study Examines How Preoperative Nutritional Status Affects Postoperative Delirium in Patients Undergoing Major Abdominal Surgery for Gynecological and Gastrointestinal Tumors. the Study Highlights the Critical Role of Preoperative Malnutrition in Delirium and Recommends That All Patients Scheduled for Major Abdominal Surgery Be Evaluated for Nutritional Status At the Outset.
Brief Title: Malnutrition is a Severe Health Issue for Cancer Patients. This Study Examines How Preoperative Nutritional Status Affects Postoperative Delirium in Patients Undergoing Major Abdominal Surgery for Gynecological and Gastrointestinal Tumors.
Status: Completed | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ozlem Sen, Anesthesiology and Reanimation Specialist MD., Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Other Study IDs: Hazel06
Record Dates: First submitted 2024-08-27; First posted 2024-10-24 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-08

CONDITIONS: Surgery; Malnutrition; Delirium, Postoperative; Abdominal Neoplasm
MeSH Terms: conditions — Malnutrition; Emergence Delirium; Abdominal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Major Abdominal Surgery — Patients with ASA I-IV, over 18 years of age, undergoing major abdominal surgery, have gynecological and GIS tumor, expected to stay in postoperative care unit for more than 24 hours.

SUMMARY:
The World Health Organization (WHO) identifies malnutrition as a significant public health threat. It is a common issue among cancer patients due to various factors. Specific nutrient deficiencies can lead to severe cognitive problems. This study aims to evaluate the impact of preoperative nutritional status on the frequency of postoperative delirium. Additionally, we will compare different parameters that can be used to diagnose preoperative malnutrition.

We included a total of 120 patients aged over 18 years, classified as ASA I-IV, who were undergoing major abdominal surgery for gynecological or gastrointestinal tumors and were expected to remain in the postoperative care unit for more than 24 hours. The patients' preoperative scores, albumin levels, prealbumin levels, and other relevant data were recorded. In the first 24 hours post-surgery, delirium was assessed using the Ramsay Sedation Scale and the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU).

ELIGIBILITY:
Inclusion Criteria:

* ASA I-IV
* Over 18 years of age
* Undergoing major abdominal surgery for gynecological and GIS tumor
* Expected to stay in postoperative care unit for more than 24 hours

Exclusion Criteria:

* Under age 18.
* Patients scheduled for emergency surgery, pregnancy, who want to withdraw from postoperative work.
* Patients with dementia, Alzheimer, psychiatric illness, illiterate people.
* Patients with speech, vision and hearing problems.
* Patients with a history of alcoholism.
* Patients who need postoperative mechanical ventilation support (patients who develop heart or respiratory failure due to COPD, heart failure, pulmonary embolism and similar reasons)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing major abdominal surgery, have gynecological and GIS tumor, expected to stay in postoperative care unit for more than 24 hours.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
CAM-ICU | 24 hours
  The confusion assessment method for the intensive care unit (CAM-ICU) is a tool used to assess delirium among patients in the intensive care unit.

CONTACTS AND LOCATIONS:
Locations (1):
- Ozlem Sen, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided